CLINICAL TRIAL: NCT01170169
Title: A Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover Bioequivalence Study to Compare Omeprazole 40 mg DR Capsules Dr. Reddy's Laboratories Ltd.,With Prilosec® 40 mg Merck & Co.Inc., USA Under Fasting Conditions
Brief Title: Omeprazole Delayed Release (DR) Capsules Bioequivalence Study of Dr. Reddys Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Assistant manager - Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 7566/05-06
Record Dates: First submitted 2010-05-31; First posted 2010-07-27 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole (Experimental): Omeprazole Delayed Release Capsules of Dr. Reddy's laboratories limited
  Interventions: Drug: Omeprazole
- Prilosec (Active Comparator): Prilosec® 40 mg of Merck & Co.Inc.
  Interventions: Drug: Prilosec

INTERVENTIONS:
Drug: Omeprazole — Omeprazole Delayed Release Capsules 40 mg
  Other Names: Prelosec 40 mg
  Arms: Omeprazole
Drug: Prilosec — Prilosec® 40 mg of Merck & Co.Inc.
  Arms: Prilosec

SUMMARY:
This study examines the bioequivalence of Dr. Reddy's Omeprazole delayed release capsules under fasting condition.

DETAILED DESCRIPTION:
This is a randomized, two-treatment, two-period, two-sequence, single dose, crossover bioequivalence study to compare Omeprazole 40 mg Delayed Release Capsules (Dr.Reddy's Laboratories Ltd.,) with Prilosec® 40 mg (Omeprazole Delayed Release Capsules (manufactured by Merck & Co., Inc., USA) in 44 healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provided written informed consent.
* Subjects who were healthy within 18-45 years of age, weighing at least 50 kg.
* Body mass index of ≥ 18 kglm2 and ≤ 25 kg/m2, with body weight not less than 50 kg.
* Subjects with normal health as determined by medical history and physical examination performed within 15 days prior to the commencement of the study (dosing in period-I).
* Subjects with normal ECG, chest X-ray (PA view) and vital signs.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.

Test product, dose, mode of administration and batch number

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2006-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Majoj K Bose, Principal Investigator — Vimta Labs Limited, 142, IDA, Phase-II, Cherlapally, Hyderabad - India-500 051